CLINICAL TRIAL: NCT04221802
Title: A Multicentre Single Arm Observational Prospective Study to Assess Demographic Characteristics Burden of Disease PRO's in Uncontrolled, Severe Eosinophilic Asthma Patients Aged 18y or Older and Qualifying for Treatment With Benralizumab in BE
Brief Title: Patient-reported Outcomes in Real-world Use of Benralizumab in Patients With Severe Eosinophilic Asthma in Belgium
Acronym: BE-REAL
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D3250R00059
Record Dates: First submitted 2019-12-05; First posted 2020-01-09 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Severe Asthma
Keywords: Severe asthma, benralizumab, real-world, observational
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to assess health and quality of life outcomes in patients treated with benralizumab, within a Belgian Real-World setting. To prove the clinical value of benralizumab in a Real-World setting, the study will document the effect of benralizumab within a time frame of 112 weeks after initiation of treatment.

DETAILED DESCRIPTION:
The aim and objective of this single arm, prospective observational study is to provide supporting RWE on the symptom relief of asthma patients qualified for benralizumab therapy in Belgium. The PRO measures consist of the Asthma Control Questionnaire (ACQ 6) as well as Patient Global Impression of Change and Severity (PGI-C and PGI-S), healthcare resource utilization (HCRU) and treatment satisfaction (TSQM-9). In addition change in daily OCS use and rate of exacerbations after initiation of benralizumab in real-world setting will be assessed

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 years or older with physician's confirmed diagnosis of severe, uncontrolled asthma
* Asthma requiring high dose inhaled corticosteroid plus long-acting β adrenoceptor agonist as maintenance treatment
* A decreased lung function (FEV1 <80%), demonstrated by spirometry in the 12 months before initiation of treatment
* Patients need to fulfil one of the criteria:

  * at least 2 hospitalizations or ER treatments for severe asthma during last 12 months, or
  * at least 2 asthma exacerbations during last 12 months (worsening of asthma with need of systemic corticotherapy for at least 3 days for non cortico-dependent patients, and/or an ER visit and or a hospitalization),
  * or cortico-dependent (at least 6 months treatment with OCS at a daily dose of 4 mg or more of methylprednisolone or 5 mg or more of prednisolone for adults)
* Peripheral blood eosinophil count ≥300cells/μl at initiation of benralizumab treatment and in the year before.
* Obtained reimbursement for treatment with benralizumab
* Provision of signed written informed consent form (ICF) indicating that they understand the purpose of the study and procedures required for participation in the study.
* Patients must be able and willing to read and comprehend written instructions and comprehend and complete the questionnaires required by the protocol.
* Benralizumab naïve and have not previously received benralizumab prior to the start of this study.

Exclusion Criteria:

* Patients currently enrolled in an interventional clinical study in parallel (i.e. have not completed) including those with biologic treatment, will be excluded from the study except for patients who are in parallel documented in the Belgian Severe Asthma Registry (BSAR).
* Concurrent biologics for asthma are not allowed except for stable allergen immunotherapy (defined as a stable dose and regimen at the time of enrolment. Acceptable wash-out periods for other asthma biologics:
* ≥30 days from last dose of previous biologic
* Patients with other documented lung disease other than asthma and not within reimbursed label.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enrol severe asthma patients who qualify for a treatment with benralizumab according to the label and Belgian reimbursement criteria and who have received reimbursement for treatment with benralizumab
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2019-12-23 (Actual); Primary Completion 2024-05-13 (Actual); Study Completion 2024-05-13 (Actual)

PRIMARY OUTCOMES:
change in patient-reported asthma related symptoms | up to 6 months after initiation of benralizumab
  assessed with the Asthma Control Questionnaire (ACQ-6). The primary outcome variable (asthma control responder) is defined as a patient who had an at least (≥) 0.5-unit improvement in ACQ-6 score.

SECONDARY OUTCOMES:
Change in patient-reported asthma related symptoms up to 112 weeks after initiation of benralizumab in a real-world setting | up to 112 weeks after initiation of benralizumab
  assessed with the Asthma Control Questionnaire (ACQ-6). The primary outcome variable (asthma control responder) is defined as a patient who had an at least (≥) 0.5-unit improvement in ACQ-6 score.
change in daily OCS use following initiation of benralizumab in real-world setting | up to 112 weeks after initiation of benralizumab
  Percent change from baseline daily OCS dose
change in asthma status in a real-world setting | up to 112 weeks after initiation of benralizumab
  assessed with the Global Impression of Severity (PGI-S). The PGI-S score will be categorized according to the following responses post-baseline: very mild, mild, moderate, severe or very severe.
  PGI-S at baseline, week 2, 4, 8, 24, 56, 80 and 112 will be presented descriptively
Rate of exacerbations after initiation of benralizumab in a real-world setting | up to 112 weeks after initiation of benralizumab
  assessed with the Number of exacerbations
change of disease severity in a real-world setting | up to 8 weeks after initiation of benralizumab
  Assessed with the Global Impression of Change (PGI-C). The PGI-C score will be categorized according to the following responses post-baseline: much better; moderately better; a little better; about the same; a little worse; moderately worse; and much worse.
  PGI-C responder endpoint (a little better, moderately better, much better) will be summarised by visit for patients.
Healthcare resource utilization in a real-world setting | up to 112 weeks after initiation of benralizumab
  assessed with the Health Care Resource Utilization Questionnaire (HCRU). The HCRU will assess number of asthma-related ED/hospital admissions, number of visits to primary care physician or specialist, number of home visits by health care professional, number of pharmacy visits and number of work/school days lost due to asthma.
change in treatment satisfaction in a real-world setting | up to 112 weeks after initiation of benralizumab
  assessed with the Treatment Satisfaction Questionnaire for Medication (TSQM-9). The TSQM-9 domain scores range from 0 to 100 with higher scores representing higher satisfaction on that domain.
  The TSQM-9 scores will be presented descriptively by domain with a focus on efficacy and satisfaction.

OTHER OUTCOMES:
Improvement of nasal polyposis relevant health status | up to 112 weeks after initiation of benralizumab
  Nasal polyposis symptoms and sense of smell will be scored on a visual analogue scale (VAS) ranging from 0 to 10 in how bothersome they were in the past month (at baseline) or versus last visit (for all other timepoints) with 0 being not at all bothersome and 10 being extremely bothersome.
  The improvement of nasal polyposis relevant health status (symptoms and sense of smell) will be presented descriptively.
Onset of effect of treatment | up to 8 weeks after initiation of benralizumab
  Assessed with one question up to what extent they agree or disagree that, during the past week, they could tell their medication was working. Answers range from strongly agree to strongly disagree.
  Patient experience of onset of effect of treatment will be presented descriptively
safety and tolerability of benralizumab after initiation of benralizumab in real-world setting | up to 112 weeks after initiation of benralizumab
  The incidence of AEs: The total number of AEs/SAEs per patient, as well as the proportion of patients with at least one AE/SAE will be summarised

CONTACTS AND LOCATIONS:
Overall Officials: Dupont Lieve, Prof., Principal Investigator — Universitair Zienkenhuis Leuven
Locations (10):
- Belgium (10):
  - Research Site, Brussels
  - Research Site, Charleroi
  - Research Site, Edegem
  - Research Site, Erpent
  - Research Site, Kortrijk
  - Research Site, La Louvière
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Mechelen
  - Research Site, Roeselare

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3250R00059&attachmentIdentifier=4eeea4bf-4485-41b7-b4b7-0a1bd16dd7ef&fileName=D3250R00059_CSR_Synopsis.pdf&versionIdentifier=